CLINICAL TRIAL: NCT02323945
Title: Mechanisms of Intermittent Hypoxia-induced Motor Recovery in Persons With SCI
Brief Title: Effects of Breathing Mild Bouts of Low Oxygen on Limb Mobility After Spinal Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: Foundation Wings For Life (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Randy Trumbower, PT, PhD, Assistant Professor, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017P001940a; 1R01HD081274-01 (NIH)
Record Dates: First submitted 2014-11-20; First posted 2014-12-24 (Estimated); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Spinal Cord Injuries
Keywords: acute intermittent hypoxia; incomplete spinal cord injury; strength; walking; breathing
MeSH Terms: conditions — Spinal Cord Injuries; Respiratory Aspiration | interventions — Insemination, Artificial, Homologous; Walking

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- AIH/Walk (Active Comparator): Subjects with chronic, motor-incomplete SCI receive acute intermittent hypoxia (AIH) with walking practice, then AIH with strength practice and compare their efficacy on enhancing strength and/or walking performance.
  Interventions: Other: AIH; Other: Walk
- AIH/Strength (Active Comparator): Subjects with chronic, motor-incomplete SCI receive AIH with strength practice, then AIH with walking practice and compare their efficacy on enhancing strength and/or walking performance.
  Interventions: Other: AIH; Other: Strength

INTERVENTIONS:
Other: AIH — Participants will breathe intermittent low oxygen via air generators. The generators will fill reservoir bags attached to a non-rebreathing face mask. Oxygen concentration will be continuously monitored to ensure delivery of fraction of inspired oxygen (FiO2) = 0.10±0.02 (hypoxia). Participants will receive treatment on 5 consecutive days.
  Other Names: Acute Intermittent Hypoxia
Other: Walk — 30 minutes of walking practice consisting of 5 repetitions of 6-minute walks
  Arms: AIH/Walk
Other: Strength — 30 minutes of isometric ankle plantar flexion torque practice broken into 3 sets of 10 repetitions
  Arms: AIH/Strength

SUMMARY:
Accumulating evidence suggests that repeatedly breathing low oxygen levels for brief periods (termed intermittent hypoxia) is a safe and effective treatment strategy to promote meaningful functional recovery in persons with chronic spinal cord injury (SCI). The goal of the study is to understand the mechanisms by which intermittent hypoxia enhances motor function and spinal plasticity (ability of the nervous system to strengthen neural pathways based on new experiences) following SCI.

DETAILED DESCRIPTION:
Accumulating evidence suggests that repeatedly breathing low oxygen levels for brief periods (termed intermittent hypoxia) is a safe and effective treatment strategy to promote meaningful functional recovery in persons with chronic spinal cord injury. Repetitive exposure to mild hypoxia triggers a cascade of events in the spinal cord, including new protein synthesis and increased sensitivity in the circuitry necessary for breathing and walking. Recently, the investigators demonstrated that daily (5 consecutive days of) intermittent hypoxia stimulated walking enhancement in persons with chronic spinal cord injury.

Despite these exciting findings, important questions remain. First, does intermittent hypoxia improve walking recovery by increasing strength or muscle coordination or both? Understanding its mechanisms will allow us to best apply intermittent hypoxia in the clinic. Second, initial studies indicate that the beneficial effects of intermittent hypoxia are greatest when intermittent hypoxia is used just prior to task training and that the benefits are greatest for the practiced task. The investigators will explore this possibility by examining the effects of intermittent hypoxia on walking ability and force production when applied alone and when applied in combination with walking training or strength training. The investigators expect to observe the greatest improvements in walking ability in those individuals receiving intermittent hypoxia with walking training and the greatest improvements in strength in response to intermittent hypoxia with strength training. Third, studies suggest that intermittent hypoxia induces spinal plasticity by increasing the expression of a key plasticity-promoting protein, brain-derived neurotrophic factor (BDNF). Mutations in the BDNF gene have been shown to impair BDNF functionality. Thus, the investigators will also explore the impact of BDNF polymorphisms on responsiveness to intermittent hypoxia therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and 75 years (the latter to reduce likelihood of heart disease)
* Medical clearance to participate
* Lesion at or below C2 and above T12 with non-progressive etiology
* Classified as motor-incomplete with visible volitional leg movement
* Injury greater than 1 year

Exclusion Criteria:

* Concurrent severe medical illness (i.e., infection, cardiovascular disease, ossification, recurrent autonomic dysreflexia, unhealed decubiti, and history of pulmonary complications)
* Pregnant women because of the unknown affects of AIH on pregnant women and fetus
* History of seizures, brain injury, and/or epilepsy
* Undergoing concurrent physical therapy
* Diabetes
* Cirrhosis
* Caffeine and/or NSAID allergies or intolerances

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2014-10; Primary Completion 2027-08 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change in overground walking endurance | Baseline, immediately after intervention (day 1 and day 5), and at follow-ups (one week and two weeks)
  Endurance will be measured as the distance walked during 2 min and 6 min (6MWT).
Change in muscle strength | Baseline, immediately after intervention (day 1 and day 5), and at follow-ups (one week and two weeks)
  Strength will be assessed as the maximum isometric torque produced by the ankle and measured by a 6 degrees-of-freedom (DOF) load cell.

SECONDARY OUTCOMES:
Change in overground walking speed | Baseline, immediately after intervention (day 1 and day 5), and at follow-ups (one week and two weeks)
  Speed will be assessed by the time required to walk 10 meters (10MWT).

CONTACTS AND LOCATIONS:
Overall Officials: Randy D Trumbower, PT, PhD, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (1):
- Spaulding Rehabilitation Hospital, Cambridge, Massachusetts, United States

REFERENCES:
- [Background] Hayes HB, Jayaraman A, Herrmann M, Mitchell GS, Rymer WZ, Trumbower RD. Daily intermittent hypoxia enhances walking after chronic spinal cord injury: a randomized trial. Neurology. 2014 Jan 14;82(2):104-13. doi: 10.1212/01.WNL.0000437416.34298.43. Epub 2013 Nov 27. PMID 24285617
- [Background] Trumbower RD, Jayaraman A, Mitchell GS, Rymer WZ. Exposure to acute intermittent hypoxia augments somatic motor function in humans with incomplete spinal cord injury. Neurorehabil Neural Repair. 2012 Feb;26(2):163-72. doi: 10.1177/1545968311412055. Epub 2011 Aug 5. PMID 21821826
- [Background] Hoffman MS, Golder FJ, Mahamed S, Mitchell GS. Spinal adenosine A2(A) receptor inhibition enhances phrenic long term facilitation following acute intermittent hypoxia. J Physiol. 2010 Jan 1;588(Pt 1):255-66. doi: 10.1113/jphysiol.2009.180075. Epub 2009 Nov 9. PMID 19900961
- [Background] Baker-Herman TL, Fuller DD, Bavis RW, Zabka AG, Golder FJ, Doperalski NJ, Johnson RA, Watters JJ, Mitchell GS. BDNF is necessary and sufficient for spinal respiratory plasticity following intermittent hypoxia. Nat Neurosci. 2004 Jan;7(1):48-55. doi: 10.1038/nn1166. Epub 2003 Dec 14. PMID 14699417
- [Background] Hayes HB, Chvatal SA, French MA, Ting LH, Trumbower RD. Neuromuscular constraints on muscle coordination during overground walking in persons with chronic incomplete spinal cord injury. Clin Neurophysiol. 2014 Oct;125(10):2024-35. doi: 10.1016/j.clinph.2014.02.001. Epub 2014 Feb 14. PMID 24618214